CLINICAL TRIAL: NCT01054963
Title: Peer to Peer Mentoring: Facilitating Individuals With Early Inflammatory Arthritis to Manage Their Arthritis - Peer Mentor Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Arthritis Network (Network)
Responsible Party: Principal Investigator, Dr. Mary Bell, Rheumatologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Purpose: Supportive Care
Other Study IDs: 419-2009
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Early Inflammatory Arthritis; Chronic Disease
Keywords: early inflammatory arthritis; chronic disease; peer support; peer mentor; peer counselling
MeSH Terms: conditions — Arthritis; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: peer mentor training — A quasi-experimental, before and after study design is proposed to obtain data for planning and implementing a larger-scale study. A training workshop for individuals with IA to become peer mentors will increase peer mentors' confidence and skills to provide one-on-one support to individuals with EIA. Using a combination of lectures, experiential learning and question/answer sessions, peer mentors will learn and practice informational, emotional, appraisal support techniques and skills (communication skills, problem-solving strategies, use of decision tools). Training will be conducted face-to-face, in small-group format by research team and others (2 sessions approx. 5 hours each), in a private meeting room at SHSC. Peer mentors will then provide support to individuals newly diagnosed with IA for 12 weeks (once per week) by telephone and /or face-to-face. Peer mentors will receive ongoing support from the research team (telephone, meetings).

SUMMARY:
Inflammatory arthritis (IA) is a major cause of long-term disability. Peer support may be a solution to the common problem of delayed treatment. Early peer support may result in improved use of therapy, higher self-efficacy, reduced anxiety, and improved coping in the first two years post-diagnosis. This study involves the development and testing of a peer mentor training initiative as one part of an intervention study for people with early IA (EIA). Peer mentors will be trained and assessed to provide one-on-one support (information, emotional, feedback) to individuals who have recently been diagnosed with IA. This is one part of an intervention study. The other part is called Peer to Peer Mentoring: Facilitating Individuals with Early Inflammatory Arthritis to Manage their Arthritis - Peer Mentoring Program.

ELIGIBILITY:
Inclusion Criteria:

* To become a peer mentor are:

  1. Diagnosis of IA from a physician
  2. Disease duration more than 2 years and managing well
  3. Currently using medications (DMARDS/biologics) to treat arthritis
  4. Have completed an Arthritis Self-Management Program (ASMP) provided by The Arthritis Society and/or similar program and/or have sufficient knowledge and experience with teaching or providing mentoring support to an individual living with a chronic disease
  5. Able to participate in two approximately 5-hour training workshops
  6. Able to take part in ongoing assessment/evaluation activities (self-report questionnaire, interviews, observation, study activity log)
  7. Able to commit to the duration of the research study
  8. Willing to provide ongoing one-on-one support to an individual newly diagnosed with IA
  9. 18 years of age or older
  10. Able to speak, understand, read and write English

Exclusion Criteria:

* Do not meet inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
ability to provide informational, appraisal and emotional support | 0, 3, 6 months

SECONDARY OUTCOMES:
confidence to provide informational, appraisal and emotional support | 0, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Bell, MD, FRCPC, Principal Investigator — Division of Rheumatology, Sunnybrook Health Science Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Sandhu S, Veinot P, Embuldeniya G, Brooks S, Sale J, Huang S, Zhao A, Richards D, Bell MJ. Peer-to-peer mentoring for individuals with early inflammatory arthritis: feasibility pilot. BMJ Open. 2013 Mar 1;3(3):e002267. doi: 10.1136/bmjopen-2012-002267. PMID 23457326